CLINICAL TRIAL: NCT07228949
Title: Real-World Analgesic Management of Complex Regional Pain Syndrome: An Observational Study in a Tertiary Care Setting
Brief Title: Complex Regional Pain Syndrome: Analgesic Outcome
Status: Not yet recruiting | Type: Observational
Sponsor: Ciusss de L'Est de l'Île de Montréal (Other)
Responsible Party: Principal Investigator, Veronique Brulotte, Doctor, Ciusss de L'Est de l'Île de Montréal
Other Study IDs: 2026-4071
Record Dates: First submitted 2025-11-13; First posted 2025-11-14 (Actual); Last update posted 2025-11-17 (Actual); Status verified 2025-11

CONDITIONS: Chronic Pain; Complex Regional Pain Syndrome
Keywords: Chronic Pain; complex regional pain syndrome
MeSH Terms: conditions — Chronic Pain; Complex Regional Pain Syndromes

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients who received at least one eligible analgesic intervention: Patient's treated at Maisonneuve-Rosemont Hospital Pain Management Centre for complex regional pain syndrome between January 2020 and October 2025 who received at least one eligible analgesic intervention (plexus or peripheral nerve block, sympathetic block, IV Ketamine infusion, IV Pamidronate infusion)

SUMMARY:
This retrospective observational study aims to describe the use and analyze the effectiveness of various analgesic interventions in patients diagnosed with Complex Regional Pain Syndrome (CRPS) at the Pain Management Center of Hôpital Maisonneuve-Rosemont (HMR) between January 2020 and October 2025.

Background:

Complex Regional Pain Syndrome is a chronic pain condition characterized by severe, persistent pain accompanied by sensory, vasomotor, sudomotor, and motor/trophic changes, often following trauma or surgery. Despite established diagnostic criteria (Budapest criteria), its pathophysiology remains poorly understood, and evidence-based treatments are limited. While multidisciplinary functional rehabilitation remains the cornerstone of management, various analgesic interventions are used to facilitate recovery when medications fail to adequately control pain.

Common interventions include:

* Plexus or peripheral nerve blocks (brachial or sciatic, with or without adjuvants such as dexamethasone or dexmedetomidine)
* Intravenous ketamine infusions
* Sympathetic blocks (stellate or lumbar)
* Intravenous pamidronate infusions

Although all these techniques are used in clinical practice, their relative efficacy and predictive factors for success remain unknown. Clinicians rely on experience rather than data-driven guidance to select an initial intervention. Identifying factors such as CRPS subtype or symptom duration that predict analgesic response could improve treatment efficiency and functional recovery.

Objectives:

Primary objective: To determine the frequency distribution of first-line analgesic interventions used in patients with CRPS treated at HMR's Pain Management Center.

Secondary objectives:

* To evaluate the success rate ("significant analgesia") of each intervention when used first-line.
* To assess the incidence of significant adverse effects.
* To analyze success rates according to CRPS clinical subtype (vasomotor, sensory, florid, or indeterminate) and symptom duration (<12 months, 12-18 months, >18 months).
* To determine the number of unsuccessful interventions required before achieving pain relief.

Methods:

This is a retrospective chart review including all adult patients with a CRPS diagnosis established using the Budapest criteria who received at least one eligible analgesic intervention during the study period. Data will be extracted from electronic medical records by the research team. Exclusion criteria include incomplete clinical documentation or missing information regarding the first consultation, intervention type, or analgesic outcome.

Collected variables include demographics, medications, CNESST (workers' compensation) status, PTSD diagnosis, trauma type, CRPS characteristics (affected limb, type, subtype, symptom duration), details of the first intervention (technique, dose, use of adjuvants), analgesic response, and adverse effects.

DETAILED DESCRIPTION:
STUDY MODEL Retrospective observational study in the form of a chart review. STUDIED POPULATION AND PERIOD Patients followed at the Maisonneuve-Rosemont Hospital Pain Management Center (PMC) for complex regional pain syndrome (CRPS) who received at least one analgesic intervention between January 1, 2020 and October 2025.

This period was chosen to obtain a sufficient number of patients and to best reflect current practice.

INCLUSION CRITERIA

• Patients with a diagnosis of complex regional pain syndrome as determined by the Budapest criteria and who received at least one of the following analgesic interventions: Intravenous ketamine infusion; Plexus block (infraclavicular, interscalene, axillary, popliteal sciatic) with or without adjuvant; Sympathetic block (stellate or lumbar); Intravenous pamidronate infusion. EXCLUSION CRITERIA

* Patients whose first consultation at the PMC is not digitized. Indeed, the process of digitizing handwritten clinical notes prior to the implementation of the electronic medical record (2017) is ongoing. Clinical notes prior to this date are therefore not always accessible in the computer system.
* Patients for whom the following data are incomplete or undocumented in the chart:

  * Patient's signs and symptoms at the first consultation at the Pain Management Center
  * First analgesic intervention performed
  * Analgesic success of the first intervention. OBJECTIVES Primary To determine the frequency distribution of first-line analgesic interventions among patients followed at the PMC for CRPS.

Secondary To determine the success rate of each intervention when used as first-line therapy. The success rate will be defined by the documentation of significant pain reduction that allowed improved function following the intervention.

To determine the proportion of patients who reported a significant adverse event between the day of the procedure and the first post-procedure follow-up visit for each intervention (pain increase, severe pain at puncture site, hematoma, infection, nausea/vomiting, nightmares, general malaise).

To determine the success rate of each analgesic intervention according to the clinical subtype of CRPS.

To determine the success rate of each analgesic intervention according to the duration of symptoms at the time of the first analgesic intervention (<12 months, 12-18 months, >18 months).

To determine the number of ineffective interventions received by each patient before achieving significant analgesia.

SAMPLE SIZE A sample size calculation will not be performed for this study. The PMC is a tertiary pain clinic that treats a large number of patients, and it is estimated that the chosen period will yield a sample of approximately 200 patients.

GENERAL PROCEDURE Data will be collected from digitized records in the Clinibase and Oacis clinical applications.

An initial sampling of charts will be performed in Clinibase by the planning, programming, and research department of the CIUSSS de l'Est-de-l'Île-de-Montréal. A search of the Clinibase database using the type of appointment at the Pain Management Center between January 1, 2020, and October 23, 2025, will provide the chart numbers of potentially eligible patients. The appointment types searched will include: block, ketamine infusion, pamidronate, stellate block, and lumbar sympathetic block.

Each chart will then be reviewed in Oacis to locate the first consultation note at the Pain Management Center in order to verify inclusion criteria-specifically, a diagnosis of complex regional pain syndrome as determined by the Budapest criteria. The use of an eligible analgesic intervention (plexus block, pamidronate infusion, ketamine infusion, stellate or lumbar sympathetic block) for the treatment of CRPS pain will be confirmed. The analgesic technique does not necessarily need to have been performed at the first visit to be eligible. Charts meeting the inclusion criteria will be retained for the research project and analyzed in more detail to collect the required data.

DATA COLLECTION

Patient data:

* Demographic data

  * Age
  * Sex
* Association of the chart with a worker's compensation agency (CNESST in Quebec) (yes/no) (This information will be collected because affiliation with a workers' compensation program is an independent factor for poorer response to analgesic interventions. It is therefore a confounding factor for the primary endpoint-intervention success) (Clin J Pain 1995;11:94-102);
* Patient's medication (SSRI antidepressants (yes/no), tricyclic antidepressants (yes/no), gabapentinoids (yes/no), NSAIDs (yes/no), opioids (yes/no))
* Initial trauma (fracture, sprain, surgery, stroke, other);
* Post-traumatic stress disorder (yes/no). This variable will be collected for the same reason as CNESST affiliation. A PTSD diagnosis significantly affects pain intensity and treatment response, particularly if inadequately addressed (J Pain Res 2018;11:527-36).

CRPS data:

* Upper or lower limb involvement;
* Left or right;
* Duration of symptoms at the time of first analgesic intervention (measured from the initiating event) (<12 months, 12-18 months, >18 months);
* Symptoms reported by the patient:

  * Sensory: hyperalgesia (yes/no), allodynia (yes/no)
  * Vasomotor: temperature asymmetry (yes/no), color asymmetry (yes/no), skin color change (yes/no)
  * Sudomotor: edema (yes/no), sweating change (yes/no)
  * Motor/trophic: decreased range of motion (yes/no), tremor (yes/no), weakness (yes/no), dystonia (yes/no), trophic changes in skin, nails and/or hair (yes/no).
* Signs observed by the physician:

  * Sensory: hyperalgesia (yes/no), allodynia (yes/no)
  * Vasomotor: temperature asymmetry (yes/no), color asymmetry (yes/no), skin color change (yes/no)
  * Sudomotor: edema (yes/no), sweating change (yes/no)
  * Motor/trophic: decreased range of motion (yes/no), tremor (yes/no), weakness (yes/no), dystonia (yes/no), trophic changes in skin, nails and/or hair (yes/no).
* CRPS category (type I, type II, ROS, NOS)
* CRPS subtype, as determined by the main symptom reported at the first consultation:

  * Vasomotor: predominance of vasomotor and sudomotor signs/symptoms
  * Sensory: predominance of sensory signs/symptoms (hyperalgesia, allodynia)
  * Florid: most symptoms present and/or motor symptoms predominant
  * Undetermined (chart notes do not allow subtype determination)

First intervention performed:

* Plexus block

  * Infraclavicular, axillary, interscalene, popliteal sciatic
  * Dose of agent used (mL)
  * Adjuvant (yes/no)
  * Type of adjuvant: dexamethasone (yes/no), dexmedetomidine (yes/no)
* Sympathetic block

  * Stellate, lumbar
  * Ultrasound-guided (yes/no), fluoroscopy (yes/no), anatomical landmarks (yes/no)
  * Dose of agent used (mL)
* Ketamine infusion

  * Dose (mg)
  * Duration (min)
  * Concomitant use of midazolam (yes/no) If yes, dose (mg)
* Pamidronate infusion o Dose (mg)

Follow-up visit data:

* Analgesic success (yes/no), defined as significant pain reduction that allowed improved function, according to patient report.
* Report of adverse effects (yes/no)
* Type of adverse effect reported: pain increase, severe pain at puncture site, hematoma, infection, nausea/vomiting, nightmares, general malaise, other)

Data from other follow-up visits:

* Number of different analgesic interventions required to achieve significant relief: 1, 2, 3, 4, or no analgesia
* Type of intervention that was beneficial (if the first intervention did not provide relief) STATISTICAL ANALYSES Data will be stored in an Excel file and analyzed with SPSS Statistics software. Continuous data will be analyzed using the Shapiro-Wilk test to assess normality. Normally and non-normally distributed values will be reported as mean (standard deviation) and median (interquartile range), respectively. Categorical data will be reported as number (percentage). The primary objective-the frequency distribution of first-line analgesic interventions-will be reported as number (percentage), as will the analgesic success rate for each intervention. The success rate of each technique by CRPS subtype and symptom duration will then be analyzed using the Chi-square or Fisher's exact test. A p < 0.05 will be considered statistically significant.

To better compare the different techniques, a propensity score approach will be used. The probability of receiving each treatment will be calculated based on the following characteristics: age, sex, symptom duration, limb type, CNESST affiliation, medications used, treating physician, and CRPS subgroup. These probabilities will be calculated using multinomial logistic regression and will define the propensity scores. Each patient's characteristics will be weighted using the Inverse Probability of Treatment Weighting (IPTW) method. After weighting, group balance will be verified by ensuring that standardized mean differences (SMD) for each covariate are below 0.1. Finally, the weighted success rate for each technique will be calculated. Weighted Odds Ratios (OR) with 95% confidence intervals will also be computed using weighted logistic regression for each treatment compared to the reference treatment. Sensitivity analyses will be performed using other weighting methods such as Overlap Weighting, 1:1 Matching, and Entropy Balancing.

To identify the best treatment for each subgroup, the probability of success as a function of treatment, subgroup, and a "treatment × subgroup" interaction term will be calculated using logistic regression. If the interaction term is significantly associated with the probability of success, stratified analyses will be conducted by subgroup. For each subgroup, a propensity score will be calculated using the same method described above, excluding the subgroup variable from adjustment. Weighted success probabilities will be calculated for each treatment and each subgroup, as well as ORs with 95% CIs compared to the reference treatment, to identify the optimal treatment for each subgroup.

ELIGIBILITY:
Inclusion Criteria:

* Patients with a diagnosis of complexe regional pain syndrome
* Patients who received at least one of the following intervention: peripheral nerve block (infraclavicular, intrerscalene, axillary, popliteal sciatic), sympathetic block (stellate, lumbar), intravenous ketamine infusion, or intravenous pamidronate infusion)

Exclusion Criteria:

* First consultation is not digitalized
* Information on signs and symptoms at the first consultation is missing

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Adult patients treated at HMR's Pain management centre for CRPS between January 1st 2020 and October 2025.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2025-11 (Estimated); Primary Completion 2026-05 (Estimated); Study Completion 2026-05 (Estimated)

PRIMARY OUTCOMES:
Frequency distribution of first-line analgesic interventions | within 6 months of first visit at the Pain Clinic
  To determine the frequency distribution of first-line analgesic interventions used in patients with complex regional pain syndrome

CONTACTS AND LOCATIONS:
Overall Officials: Veronique Brulotte, MD, Principal Investigator — CIUSSS-de-l'Est-de-l'Ile-de-Montréal
Locations (2):
- Canada (2):
  - Maisonneuve-Rosemont Hospital, Montreal, Quebec
  - Hopital Maisonneuve Rosemont, Montreal

IPD SHARING:
Plan to Share IPD: No